CLINICAL TRIAL: NCT02961205
Title: Nutrition Supplementation in Cardiovascular Surgery Patients-A Randomized Controlled Pilot Trial
Brief Title: Nutrition Supplementation in Cardiovascular Surgery Patients
Acronym: NutriSuP-CVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INN16-003
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Nutritional Supplementation (Experimental): Patients randomized to the interventional arm will receive Ensure Enlive (Abbott Nutrition), a high energy, high protein oral supplement.
  Interventions: Dietary Supplement: Oral Nutritional Supplementation
- Standard of care (No Intervention): Patients randomized to the control arm will continue their usual diet.

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplementation — Participants randomized to this arm will receive one bottle of Ensure Enlive 2 times per day, for 30 days prior to their cardiovascular surgery, plus continue their usual diet.
  After their CVS and throughout their hospitalization they will continue to receive 2 bottles of Ensure Enlive per day, plus the standard hospital menu (3 meals per day, plus snacks or as ordered by the medical team), ending at hospital discharge.
  Other Names: Ensure Enlive
  Arms: Oral Nutritional Supplementation

SUMMARY:
This randomized controlled pilot study evaluates the use of oral nutritional supplementation in nutritionally at-risk cardiovascular surgery patients. The oral nutrition supplement is given for 30 days prior to surgery, continuing throughout their surgical hospitalization and ends at hospital discharge. Half of the participants will receive the oral nutritional supplement and the other half will not.

DETAILED DESCRIPTION:
Cardiovascular surgery (CVS) is a resource intensive modality in the treatment of coronary artery disease and valvular heart disease. CVS patients who are malnourished experience increased duration of cardiopulmonary bypass, post-operative infections, impaired wound healing, muscle wasting, longer lengths of intensive care unit (ICU) and hospital stay, higher readmission rates, higher treatment costs and marked increases in mortality. Despite the devastating effects of malnutrition in these patients, physicians and health care practitioners are poor in respect to identification, monitoring and treatment of malnutrition.

In two large tertiary hospitals in Ontario, this will be a randomized trial of a novel nutritional pathway to rapidly identify at-risk CVS patients pre-operatively, and then provide oral nutritional supplementation (ONS) during the 30 days prior to surgery, then continue supplementation throughout hospitalization until discharge. Meaningful patient-centered and economic outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Require cardiovascular surgery
2. Have been assessed in a pre-operative clinic
3. Have an intermediate or high risk Society of Thoracic Surgeons (STS) score
4. Malnutrition Universal Screening Tool (MUST) score of >1.

Exclusion Criteria:

1. Require urgent/emergent cardiovascular surgery
2. Have advanced symptomatic angina or heart failure
3. Are designated palliative care
4. Are currently suffering from refeeding syndrome
5. Have a pre-existing medical condition that prevents oral intake of full fluids
6. Are on a fluid restricted diet
7. Are unable to walk prior to current illness
8. Have a current diagnosis of diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome
9. Are pregnant or currently breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Recruitment | 1 year
  This pilot study will be considered as successfully demonstrating feasibility of recruitment if 60 participants are recruited over 12 months. The overarching objective of this pilot study is to prove feasibility of recruitment and of the protocol in order to continue to a large phase 3 trial.

SECONDARY OUTCOMES:
Nutrition Status | 30 days post surgery date
  The Malnutrition Universal Screening Tool (MUST) will be the method of assessment. The MUST is a five-step screening tool to identify adults, who are at-risk of malnutrition.
Functional Performance | 30 days post surgery date
  Six Minute Walk Test will be the method of assessing physical function and therapeutic response to the intervention. Patients will be asked to walk as far as possible in six minutes, going at their own pace and resting as needed, along a marked walkway.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rahman, MD FRCPC, Principal Investigator — St. Joseph's Health Care, London ON
Locations (1):
- LHSC-University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No